CLINICAL TRIAL: NCT06380335
Title: A Multicentre, Observational Study in Patients With Liver Cirrhosis Who Have Hepatic Decompensation (OPAL)
Brief Title: Study in Patients With Decompensated Liver Cirrhosis
Acronym: OPAL
Status: Active, not recruiting | Type: Observational
Sponsor: Resolution Therapeutics Limited (Network)
Responsible Party: Sponsor
Other Study IDs: RTX001-01S
Record Dates: First submitted 2024-04-09; First posted 2024-04-23 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Liver Cirrhosis
Keywords: Liver cirrhosis; Cirrhotic; Hepatic Cirrhosis; Chronic Liver Disease; Liver Fibrosis; Decompensated liver cirrhosis; Child-Pugh Score; MELD score; Liver function tests; Hepatic encephalopathy; End Stage Liver Disease (ESLD); Retractable ascites; Variceal Bleeding
MeSH Terms: conditions — Liver Cirrhosis; Hepatic Encephalopathy; End Stage Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients with liver cirrhosis who have been hospitalised following a recent hepatic decompensation which is at least 6 months after any hospitalisation for a prior decompensation event.
- Group 2: Out-patients with medically refractory ascites that recurs (i.e., second LVP) within a 6-month period.

SUMMARY:
OPAL is a multicenter observational study, following the natural disease trajectory of participants who have permanent damage to their liver caused by scarring, sometimes also referred to as liver cirrhosis. These participants will also have recently had an acute worsening of their liver disease, which is also known as a hepatic decompensating event, which has resulted in them being admitted to hospital or required them to seek medical attention as an outpatient.

DETAILED DESCRIPTION:
This multicenter, observational natural history study is designed to follow the disease trajectory of adults with cirrhosis of the liver who have a qualifying hepatic decompensation event.

The primary objective of the study is to obtain real world data to understand the clinical course of cirrhotic patients following a decompensation event in order to generate data to provide context for the safety and efficacy evaluation of future interventional treatments. Observed data will be collected from the visits and assessments conducted as part of the routine standard of care (SOC) follow-up of these patients. In addition, given the variability in SOC and timing of follow-up visits across institutions, if study required assessments do not coincide with a routine SOC visit at the institution, blood draws and other study-specific assessments will be collected at defined time points for the study analysis.

All participants who meet the eligibility criteria and stabilize following a hepatic decompensation event will have their clinical course followed for up to 96 weeks, and then be invited to participate in the study long term follow observational phase for a further 3 years.

ELIGIBILITY:
Individuals eligible to participate in this study must meet the following criteria:

Inclusion Criteria:

1. Male or female age ≥18-75 years.
2. Patient is willing and able to provide informed consent to participate in the study.
3. Patient confirms willingness/ability to comply with all study procedures.
4. Has a diagnosis of liver cirrhosis determined by a physician based on at least one of the following:

   1. clinical and radiological features that correlate with a diagnosis of cirrhosis;
   2. transient elastography (TE) (FibroscanTM) >15kPa;
   3. previous liver biopsy confirming histological features of cirrhosis.
5. 5. For eligibility at Screen Part 2 - Aetiology of liver disease of steatotic liver disease (SLD) including pure metabolic dysfunction associated steatotic liver disease (MASLD) or metabolic and alcohol related/associated liver disease (Met-ALD), or alcohol-related liver diseases (ALD).

   a. Patients with ALD or Met-ALD only if they are confirmed to not be drinking alcohol above Met-ALD limits defined in this protocol AND have phosphatidyl ethanol (PEth) test <200 ng/ml. (N.B. No more than 34% of the total patients in this protocol will be ALD [excludes Met-ALD]).
6. Meets one of the following criteria:

   1. a. Hospitalised as an in-patient for a recent major hepatic decompensation event (qualifying event) including ascites, HE or variceal bleed, HRS-AKI or SBP, this being the only hospitalisation for an hepatic decompensation event within the last 6 months, and where recent is defined as within 6 weeks of hospital discharge OR
   2. Out-patient: Medically refractory ascites is defined by the repeated (≥ 2) need for LVP (i.e., therapeutic, not diagnostic) at least once per 8 weeks despite best medical attempts to control the ascites by sodium restriction and diuretic treatment, as confirmed by the Investigator, with date on of onset [defined as the date of the second therapeutic paracentesis] occurring within the past 6 months.
7. MELD 3.0 score of 12-20 taken within 2 weeks of qualifying event.
8. Has stabilised post-hepatic decompensation event, as defined by two MELD assessments (within 1 point of each) other taken within 2 weeks, or physician assessed as stable. with the ability to safely cell mobilise with GCSF, apherese and received RTX001 treat in the interventional Phase 1/2 study.

Exclusion Criteria:

1. Liver cirrhosis due to:

   1. any viral hepatitis , or
   2. autoimmune and cholestatic aetiologies including, but not limited to, primary biliary cholangitis and primary sclerosing cholangitis.
2. Acute liver disease in the absence of underlying liver cirrhosis, including, but not limited to, drug induced liver injury.
3. Any current organ failure requiring more than out-patient non-invasive supportive care, and not associated with the patient's qualifying hepatic decompensation event.
4. Known splenomegaly ≥16cm.
5. Thrombocytopenia <50,000 mm3.
6. Sepsis (with positive microbial cultures) or as defined by the Investigator, unless stable and is at least 4 weeks after having completed a full course of intravenous antibiotics.
7. Presence or suspicion of any of the following co-morbidities:

   1. a. history of liver transplantation or other organ transplant;
   2. ACLF;
   3. known human immunodeficiency virus;
   4. pulmonary embolism;
   5. hepatocellular carcinoma, or active malignant disease within the last 5 years, (excluding non-melanoma skin cancer, cervical carcinoma in situ, superficial bladder cancer, benign polyps etc.);
   6. co-hepatic morbidities e.g., portal vein thrombosis;
   7. hepatic hydrothorax unless it is a small hydrothorax, not clinically apparent, that is detected incidentally by radiologic evaluation that does not require clinical intervention.
   8. chronic renal impairment (on dialysis) or unresolved acute kidney injury;
   9. acute or chronic heart failure (New York Heart Association Grade III/IV);
   10. porto-pulmonary hypertension;
   11. severe chronic lung disease e.g., chronic obstructive pulmonary disease or interstitial lung disease where the forced expiratory volume (FEV1) is less than 50% and/or FEV1/forced vital capacity is less than 60%;
   12. hepatopulmonary syndrome;
   13. history or current treatment with chronic albumin treatment;
   14. significant untreated/unstable psychiatric disease;
   15. transjugular intrahepatic portosystemic shunt (TIPSS) within the previous 6 months.
8. Current or planned use of immunosuppressive medication, with the exception of low doses up to 10 mg/day prednisone or equivalent, or inhaled steroids to manage an asthma, which are permitted.
9. Any other intercurrent illness that is either life-threatening or of clinical significance such that it might limit compliance with study procedures, in the Investigator's opinion.
10. Current alcohol misuse defined as alcohol intake greater than 3 units/day for females and 4 units/day for males, or binge drinking (>14 units/day) as determined by the Investigator or PEth alcohol test >200 ng/ml. One alcohol unit is equivalent to14 g of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits. Note: patients with history of exceeding these alcohol use limits, if meeting all other inclusion/exclusion criteria, are limited to 34% of enrolled patients.
11. Intake of non-medically supervised drugs of abuse that is judged (by the Investigator) to be a high risk to the patient's acute health or which makes the patient likely to be non-compliant with follow-up.
12. Are currently participating in an investigational interventional study. Note: concurrent participation in another non-interventional study is permitted.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with liver cirrhosis who have been hospitalized for hepatic decompensation.
  2. Out-patients with refractory ascites that does not require in-patient admission.
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2030-04-03 (Estimated); Study Completion 2030-04-03 (Estimated)

PRIMARY OUTCOMES:
Examine the characteristics of patients admitted to hospital with hepatic decompensation. | Baseline and up to 96 weeks
  Demographics
Examine the characteristics of patients admitted to hospital with hepatic decompensation. | Baseline and up to 96 weeks
  Aetiology of liver disease
Examine the characteristics of patients admitted to hospital with hepatic decompensation. | Baseline and up to 96 weeks
  Disease co-morbidities
Examine the characteristics of patients admitted to hospital with hepatic decompensation. | Baseline, and up to 96 weeks
  Alcohol use
Examine the characteristics of patients admitted to hospital with hepatic decompensation. | Baseline, and up to 96 weeks
  Changes in Model for End-Stage Liver Disease (MELD) score
Examine the characteristics of patients admitted to hospital with hepatic decompensation. | Baseline, and up to 96 weeks
  Safety laboratory (biochemistry and haematology) parameters

SECONDARY OUTCOMES:
Follow the natural history of patients admitted to hospital with hepatic decompensation. | Screening up to 96 weeks
  Death or liver transplantation
Follow the natural history of patients admitted to hospital with hepatic decompensation. | Screening up to 96 weeks
  Major hepatic decompensation events
Follow the natural history of patients admitted to hospital with hepatic decompensation. | Screening up to 96 weeks
  Hospitalisations or intensive care unit (ICU) admissions
Follow the natural history of patients admitted to hospital with hepatic decompensation. | Screening up to 96 weeks
  Changes in Model for End-Stage Liver Disease (MELD) score
Examine the characteristics and natural history of patients with medically refractory ascites that do not require hospitalisation. | Screening up to 96 weeks
  Demographics
Examine the characteristics and natural history of patients with medically refractory ascites that do not require hospitalisation. | Screening up to 96 weeks
  Safety laboratory (biochemistry and haematology) parameters
Examine the characteristics and natural history of patients with medically refractory ascites that do not require hospitalisation. | Screening up to 96 weeks
  Disease co morbidities
Examine the characteristics and natural history of patients with medically refractory ascites that do not require hospitalisation. | Screening up to 96 weeks
  Alcohol use
Examine the characteristics and natural history of patients with medically refractory ascites that do not require hospitalisation. | Screening up to 96 weeks
  Changes in MELD score
Examine the characteristics and natural history of patients with medically refractory ascites that do not require hospitalisation. | Screening up to 96 weeks
  Death or liver transplantation
Examine the characteristics and natural history of patients with medically refractory ascites that do not require hospitalisation. | Screening up to 96 weeks
  Further hepatic decompensation events

OTHER OUTCOMES:
Explore clinical and laboratory parameters. | Screening up to 96 weeks
  Common clinical laboratory parameters to assess end stage liver disease.
Evaluate the effect of disease progression on biomarkers of inflammatory activity | Screening up to 96 weeks
  Additional non-invasive biomarkers of liver fibrogenesis or fibrolysis and/or molecules reflecting hepatic function.

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (2):
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital General Universitario Gregorio Marañón, Madrid
- United Kingdom (10):
  - Bristol Royal Infirmary, Bristol
  - Royal Infirmary Edinburgh, Edinburgh
  - Leeds Teaching Hospital NHS Trust, Leeds
  - Royal Liverpool Hospital, Liverpool
  - King's College Hospital, London
  - St George's Hospital, London
  - St Mary's Hospital, London
  - Nottingham University Hospital, Nottingham
  - Southampton General Hospital, Southampton
  - Sunderland Royal Hospital, Sunderland

IPD SHARING:
Plan to Share IPD: Undecided